CLINICAL TRIAL: NCT02494700
Title: Ultra Low Dose 4 Gy Orbital Radiation for Definitive Therapy of Indolent B Cell Lymphoma
Brief Title: Ultra Low Dose Orbital Radiation Therapy in Treating Patients With Stage I-IV Indolent B-cell Lymphoma or Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1046; NCI-2015-01203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-1046 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Ann Arbor Stage I B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage I Grade 1 Follicular Lymphoma; Ann Arbor Stage I Grade 2 Follicular Lymphoma; Ann Arbor Stage I Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage I Mantle Cell Lymphoma; Ann Arbor Stage II B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage II Grade 1 Follicular Lymphoma; Ann Arbor Stage II Grade 2 Follicular Lymphoma; Ann Arbor Stage II Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage II Mantle Cell Lymphoma; Ann Arbor Stage III B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage III Grade 1 Follicular Lymphoma; Ann Arbor Stage III Grade 2 Follicular Lymphoma; Ann Arbor Stage III Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage III Mantle Cell Lymphoma; Ann Arbor Stage IV B-Cell Non-Hodgkin Lymphoma; Ann Arbor Stage IV Grade 1 Follicular Lymphoma; Ann Arbor Stage IV Grade 2 Follicular Lymphoma; Ann Arbor Stage IV Indolent Adult Non-Hodgkin Lymphoma; Ann Arbor Stage IV Mantle Cell Lymphoma; Ocular Adnexal Lymphoma; Ocular Adnexal Mucosa-Associated Lymphoid Tissue Lymphoma; Orbit Lymphoma
MeSH Terms: conditions — Orbital lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (low dose orbital EBRT) (Experimental): Patients undergo two fractions of low dose orbital EBRT on 2 consecutive days. Patients experiencing stable or progressive disease after 12-16 weeks of EBRT undergo additional low dose orbital EBRT over 10 fractions. Patients experiencing partial response or minimal response 1 year after EBRT also undergo low dose orbital EBRT over 10 fractions.
  Interventions: Radiation: External Beam Radiation Therapy; Drug: Orbital Radiation

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo orbital EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation
Drug: Orbital Radiation — Participants receive radiation to entire involved orbit for a total dose of 4 Gy in 2 fractions over two consecutive days with external beam radiotherapy. If there is stable disease or progressive disease, an additional 20 Gy administered to involved site. If there are two consecutive evaluations with no change in disease burden then an additional 20 Gy administered. At one year if there is persistent disease, an additional 20 Gy administered to involved site.
  Other Names: XRT

SUMMARY:
This phase II trial studies how well ultra low dose orbital radiation therapy works in treating patients with stage I-IV low grade (indolent) B-cell lymphoma or mantle cell lymphoma involving the orbit of the eye (space enclosed by the borders of the eye socket). Orbital radiation therapy uses external beam radiation to destroy cancer cells. Using ultra low dose orbital radiation therapy may be effective in treating indolent B-cell lymphoma or mantle cell lymphoma involving the eye and may have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of ultra low dose 4 Gray (Gy) orbital radiation, measured as local orbital control (i.e. local control within the radiation field), in patients with limited and advanced stage low grade B lymphocyte (B cell) lymphoma and mantle cell lymphoma involving the ocular adnexa.

II. To evaluate the efficacy of ultra low dose 4 Gy orbital radiation, measured as complete response, in patients with limited and advanced stage low grade B cell lymphoma and mantle cell lymphoma involving the ocular adnexa.

III. To evaluate the acute and chronic toxicity of radiation to the orbit.

SECONDARY OBJECTIVE:

I. To determine if dynamic contrast enhanced magnetic resonance imaging can predict response to ultra low dose radiation therapy.

OUTLINE:

Patients undergo low dose orbital external beam radiation therapy (EBRT) on 2 consecutive days. Patients experiencing stable or progressive disease after 12-16 weeks of EBRT undergo additional low dose orbital EBRT over 10 fractions. Patients experiencing partial response or minimal response 1 year after EBRT also undergo low dose orbital EBRT over 10 fractions.

After completion of study treatment, patients are followed up every 3-4 months for 6-8 months, every 6-12 months for up to 2 years, and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with stage I-IV indolent B cell lymphoma, including MALT and follicular grade I/II. Patients with mantle cell lymphoma will also be included in this study, as mantle cell lymphoma is also radiosensitive, despite it not being an indolent B cell lymphoma. Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) are ineligible.
* Patients must have measurable disease within the orbit, either clinically and/or radiographically after biopsy confirmation of B cell lymphoma.
* Bilateral ocular adnexal involvement is permitted, if biopsy confirms unilateral disease and there is high clinical suspicion for bilateral disease, biopsy of the contralateral ocular adnexa can be waived.
* Female patients of childbearing potential must have a negative serum pregnancy test (βhCG) within 2 weeks of protocol entry.
* Planned systemic therapy after orbital radiation therapy is permitted however the timing of systemic therapy will be recorded and patients will be stratified according to receipt of adjuvant systemic therapy.
* Male patients must agree to use a barrier method of contraception or agree to abstain from heterosexual activity for the duration of the study.
* Female patients must be willing to use two adequate barrier methods of contraception to prevent pregnancy or agree to abstain from heterosexual activity throughout the study or be post-menopausal (free from menses > two years or surgically sterilized).
* Patients must have the ability to give informed consent.

Exclusion Criteria:

* Patients treated with chemotherapy for lymphoma within 4 weeks of protocol enrollment (including Rituxan).
* Patients with aggressive B cell lymphoma histology, including diffuse large B cell lymphoma (DLBCL) and grade 3 follicular lymphoma.
* Patients with chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL).
* Patients with a history of prior radiation to the orbit if re-treatment would exceed known orbital tolerance.
* Patients with pre-existing retinopathy.
* Patients who are pregnant.
* Patients with active lupus or scleroderma are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Local orbital control (i.e. local control within the radiation field) | Up to 2 years post-radiation
  Local orbital event will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Complete response rate | Up to 2 years
  Response rate will be estimated along with 95% confidence intervals.
Local regional control (i.e. local control within the ipsilateral orbit but outside of the radiation field) | Up to 2 years post-radiation therapy
Overall survival (OS) | Up to 2 years
  OS will be estimated using the Kaplan-Meier method.
Freedom from distant relapse rates | Up to 2 years
Incidence of acute and chronic ocular toxicities graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 2 years
  Toxicity data will be summarized by frequency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsea C Pinnix, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pinnix CC, Dabaja BS, Gunther JR, Fang PQ, Wu SY, Nastoupil LJ, Strati P, Nair R, Ahmed S, Steiner R, Westin J, Neelapu S, Rodriguez MA, Lee HJ, Wang M, Flowers C, Feng L, Esmaeli B. Response-Adapted Ultralow-Dose Radiation Therapy for Orbital Indolent B-Cell Lymphoma: A Phase 2 Nonrandomized Controlled Trial. JAMA Oncol. 2024 Sep 1;10(9):1195-1203. doi: 10.1001/jamaoncol.2024.2112. PMID 38990564
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org